CLINICAL TRIAL: NCT06906211
Title: Low Intensity Focused Ultrasound for Chronic Pain: High Resolution Targeting of The Human Insula
Acronym: LIFU_Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Washington D.C. Veterans Affairs Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 1781312
Record Dates: First submitted 2025-02-13; First posted 2025-04-02 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-01

CONDITIONS: Chronic Back Pain; Chronic Pain (Back / Neck)
Keywords: low intensity focused ultrasound; chronic back pain; chronic pain; functional magnetic resonance imaging
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Intervention Model Description: within-subject, randomized, double-blind, sham-controlled trial
Who Masked: Participant, Investigator
Masking Description: The Sham condition will be conducted using an interface which does not allow ultrasound energy to pass from the transducer to the target. The administration of LIFU/sham will be conducted in a double-blind fashion.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- LIFU/Sham (Other): double-blind, sham-controlled, crossover study in N=66 individuals with Chronic Back Pain
  Interventions: Device: low intensity focused ultrasound (LIFU)
- Sham/LIFU (Other): double-blind, sham-controlled, crossover study in N=66 individuals with Chronic Back Pain
  Interventions: Device: low intensity focused ultrasound (LIFU)

INTERVENTIONS:
Device: low intensity focused ultrasound (LIFU) — Low-intensity focused ultrasound (LIFU) provides an energy source with millimeter resolution that can be focused anywhere in the brain safely and effectively for non-invasive and transient neuromodulation. LIFU is an important advance and of great significance for brain-mapping efforts, diagnostics, and therapies in neuroscience and particularly promising for addiction therapy as it provides unprecedented non-surgical access to the brain regardless of depth. Much lower intensities of focused ultrasound (LIFU) are used so that tissue damage does not occur, but neural activity can be modulated. LIFU utilizes acoustic energy at much lower levels to affect tissue by mechanical effects.

SUMMARY:
In this study, the research team will use low-intensity focused ultrasound (LIFU) to temporarily change brain activity in a brain region that is known to be involved in chronic pain. Through this, the research team hopes to learn about how the brain area works in response to pain. There are main questions this study aims to answer:

* The effect of LIFU to inhibit the posterior region of the insula (PI) compared to sham stimulation in individuals with chronic back pain (CBP) and widespread pain symptoms.
* The effect of LIFU to PI compared to sham stimulation to reduce pain intensity and magnitude of the Neurologic Pain Signature (NPS) in response to evoked thermal pain.
* The effect of LIFU to PI compared to sham stimulation to reduce pain intensity and magnitude of Tonic Pain Signature in response to tonic pain.

DETAILED DESCRIPTION:
Chronic pain is a major public health problem. An estimated 100 million Americans have experienced chronic pain producing significant economic and social burden. The estimated annual cost of chronic pain is as high as $635 billion. Pharmacological treatments frequently require the use of opioids resulting in a major epidemic of abuse in the United States. New, non-addicting treatments for pain are critically needed. Neuromodulation with low-intensity focused ultrasound (LIFU) could represent a non-pharmacological treatment for chronic pain. The millimeter spatial specificity of LIFU makes it a powerful alternative to both invasive neurosurgical procedures and other noninvasive brain stimulation techniques. One promising target to treat chronic pain is the insular cortex. The insula as a key brain area involved in both sensory and affective components of chronic pain, including central sensitization processes which occur with pain chronicity. The insula is inaccessible using conventional noninvasive neuromodulatory techniques like transcranial magnetic stimulation. In contrast, LIFU can be focused deeply and provides the spatial resolution to resolve individual sub-regions of the insula. This is relevant to pain as the posterior subregion of the insula (PI) receives nociceptive input from spinothalamic tracts, relays it to the anterior insula which integrates expectation, awareness, and emotion to form the overall experience of pain. Therefore, using LIFU can address a gap in knowledge regarding the causal role of insular subregions in modulating pain response and CS processes. The preliminary data indicate that LIFU to PI reduces laboratory measures of central sensitization and evoked pain in healthy controls but there was no such effect of LIFU to anterior insula. Building on these results, the overall objective of this proposal is to examine the effect of LIFU to PI on the central sensitization processes that are a key feature of chronic pain syndromes and on neural response to evoked and tonic pain/pain intensity. The investigators will employ well validated laboratory measures of central sensitization and multivariate measures of neural response to evoked (Neurologic Pain Signature, NPS) and tonic (Tonic Pain Signature) pain. The chronic pain condition that the investigators will focus on in this study will be chronic back pain (CBP) with widespread pain widespread pain as the back is the most common site of chronic pain, is significantly more likely to be severe in the veteran population, and it commonly occurs with features of central sensitization. Eligible participants will have CBP with symptoms of widespread pain.

ELIGIBILITY:
Inclusion Criteria:

* Veterans aged 21 to 75 with Chronic Back Pain (CBP).
* CBP duration daily for last 3 months or half of days for last 6 months
* Endorse pain rating of 4/10 BPI-SF
* Evidence of widespread pain symptoms as determined by report of CBP and pain in a contralateral limb (pain in the upper, lower, left or right side of the body) in fewer than 11 sites. Upper body sites include hand, wrist, elbow or shoulder. Lower sites include hip, knee, ankle or foot.

Exclusion Criteria:

* Surgery recommended as primary treatment intervention for CBP
* Current diagnosis of fibromyalgia
* Current substance use disorder other than nicotine.
* Psychiatric disorder and not on a stable pharmacologic regimen for ≥ 4 weeks prior to screening
* Opiate use daily
* Currently pregnant or breast feeding.
* Unable to understand the consent form.
* History of head injury with loss of consciousness for more than 5 minutes, seizures, history of stroke, brain surgery, brain tumor, multiple sclerosis.
* History of metastatic cancer, rheumatoid arthritis, polymyalgia rheumatica, scleroderma, lupus, or polymyositis
* Unintended weight loss of 20 pounds or more in the last year
* Cauda equina syndrome
* Ferromagnetic implants or other contraindications for MRI
* Uncompensated congestive heart failure, unstable angina, poorly controlled arrhythmia, active systemic infection end stage renal disease.

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2025-01-15 (Actual); Primary Completion 2028-01-26 (Estimated); Study Completion 2028-01-26 (Estimated)

PRIMARY OUTCOMES:
Measures of Central Sensitization - Thermal Pain Threshold | immediately prior to 1 session LIFU and within 1 hour post LIFU; immediately prior to 1 session sham and with in 1 hour post shamdays
  For the first measure, the probe is placed on the skin on the ventral aspect of the forearm on the nondominant arm. The temperature is set at 32°C and the temperature is increased at a rate of 1°C/s to a maximum of 52°C. Participants will be asked to press a button when the heat reaches a painful level. The outcome is the temperature at this level. Heat PT are averaged over three trials each separated by 40 seconds. Thermal PT will be performed prior to and after LIFU. On each trial, the thermode is moved to a different site on the forearm to avoid sensitization and response suppression of cutaneous heat receptors.
Measures of Central Sensitization - Temporal Summation of Pain | immediately prior to 1 session LIFU and within 1 hour post LIFU; immediately prior to 1 session sham and with in 1 hour post shamdays
  The second measure refers to the perception of increasing pain in response to repeated same noxious stimuli delivered at a frequency of > 0.33 Hz. Temporal summation of pain serves as a proxy measure of pain facilitation and CS. Individuals with enhanced temporal summation of pain have facilitated ascending nociceptive processing and reduced pain-modulatory capacities. Following the temporal summation of pain paradigm, three stimulus trains of trapezoid heat pulses of 1.5 s duration will be delivered to the dorsum of the dominant hand at an inter-pulse interval of 2.5 seconds at individual subject heat pain of 6/10 on numeric pain rating scale. A total of 5 stimuli will be delivered per train. Participants will be required to rate each stimulus (0-10). The Δ scores from 5th to 1st stimulus of each train will be averaged.
Measures of Central Sensitization - Conditioned Modulation of Pain | immediately prior to 1 session LIFU and within 1 hour post LIFU; immediately prior to 1 session sham and with in 1 hour post shamdays
  A type of counter-irritation paradigm that can be used as a proxy measure for descending anti-nociceptive or pain modulation activity. CPM involves presentation of a conditioning pain stimulus to a remote area of the body while a nociceptive (test) stimulus (TS) is applied to the contralateral (heterotopic) area. We will employ conditioned modulation of pain according to using a sequential conditioning-test stimulus protocol as recommended by. The test stimulus consists of a two-minute thermal stimulus applied with the thermode at a rating of 5/10 on the numeric pain rating scale. Participants will rate their perceived pain (0-10, numeric pain rating scale) every 15 seconds. This will be performed pre/post the conditioning stimulus. The conditioning stimulus will be a cold pressor test.. The non-dominant arm will be immersed in a cold-water bath (12°C) for two minutes. This method recruits inhibitory conditioned modulation of pain because it is a strong nociceptive stimulation.

SECONDARY OUTCOMES:
Neurologic Pain Signature | immediately prior to 1 session LIFU and within 1 hour post LIFU; immediately prior to 1 session sham and with in 1 hour post shamdays
  A secondary outcome is the pain intensity and magnitude of the NPS in response to evoked thermal pain using task-based functional magnetic resonance imaging.
Tonic Pain Signature | immediately prior to 1 session LIFU and within 1 hour post LIFU; immediately prior to 1 session sham and with in 1 hour post sham
  A secondary outcome is the pain intensity and magnitude of Tonic Pain Signature in response to tonic pain using resting-state functional magnetic resonance imaging.

CONTACTS AND LOCATIONS:
Overall Officials: Mary R Lee, MD, Principal Investigator — Washington D.C. Veterans Affairs Medical Center
Locations (1):
- Washington DC Veterans Affairs Medical Center, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: Yes
behavioral and imaging data
Supporting Information: SAP, Analytic Code
Time Frame: data will be available after analysis of primary and secondary outcomes are completed